CLINICAL TRIAL: NCT06671886
Title: Testing the Effectiveness of NAFLD Clinical Care Pathway in VA Primary Care
Brief Title: NAFLD Clinical Care Pathway
Acronym: NCCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 22-071; HX003655-01A2 (Other Grant/Funding Number: VA HSR&D)
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: NAFLD; MASLD
Keywords: NAFLD; Veterans; Primary health care; MASLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — trigger factor, E coli

STUDY DESIGN:
Intervention Model Description: The study is a cluster-randomized trial to test the effectiveness of the NCCP intervention relative to Usual Care on patient-level clinical process outcomes. The unit of randomization will be the PACT team enrolled into the NCCP or usual care. Outcome assessments will be conducted at 6 and 12 months.
Who Masked: Participant
Masking Description: PACT teams will be randomized to the intervention or control arms of the study. Patients will not be individually recruited or randomized for the cluster-randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E-trigger (Experimental): The NCCP Intervention is made up of multiple components. The investigators will start by applying the e-trigger and assessing the FIB-4 score, and then will train and educate PACT personnel on managing patients with positive triggers, including making treatment recommendations in collaboration with an inter-professional team. The e-trigger will be generated every three months.
  Interventions: Behavioral: E-trigger
- Usual care (No Intervention): The control group will receive no additional training or education. PACTs will provide usual care.

INTERVENTIONS:
Behavioral: E-trigger — The NCCP Intervention is multicomponent. First, the investigators will apply the e-trigger and calculate FIB-4, and second, will educate and train PACT personnel on how to deal with trigger positive patients as well as make treatment recommendations within an inter-professional team. The e-trigger will be generated every 3 months. The effectiveness of the trigger will be assessed using the outcomes previously mentioned.
  Arms: E-trigger

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a new condition that has become the most common chronic liver disease in the world and a main cause of liver cirrhosis, liver failure and liver cancer. Obesity and diabetes, conditions that are very common among Veterans are the main risk factors for NAFLD. Therefore, the burden of NAFLD and its complications among Veterans is substantial. However, most VA patients with NAFLD are undiagnosed and untreated, and their care is not consistent with practice guidelines. The NAFLD Clinical Care Pathway (NCCP) intervention seeks to close this major gap in the care of Veterans by automatically identifying patients at risk of NAFLD, calculating their risk scores of having severe NAFLD, and educating the primary care providers on the diagnosis and treatment of NAFLD. This clinical trial will test the benefit of this NCCP intervention against usual care in increasing the rates of NAFLD diagnosis as well as referral to and enrollment in appropriate treatment. The study will also identify barriers and promotors of future NCCP implementation.

DETAILED DESCRIPTION:
Background: In the United States, non-alcoholic fatty liver disease (NAFLD) affects 25-30% of adults and has become a leading cause of chronic liver disease including cirrhosis and liver cancer. The burden of NAFLD and its complications among patients in the Department of Veterans Affairs (VA) is increasing. Most complications occur among patients with advanced hepatic fibrosis. Treatment (e.g., weight loss) improves patients' outcomes.

Significance: The investigator's data indicate that most VA patients with NAFLD are undiagnosed and untreated. There is an urgent need to address this major gap in care. Most people with NAFLD are seen in primary care settings. The NAFLD Clinical Care Pathway (NCCP) is a multistep, algorithmic process that entails identification of patients at risk through an e-trigger (Step 1), targeted history and lab testing (Step 2), noninvasive testing for hepatic fibrosis using FIB-4 (Step 3), elective additional fibrosis testing with Fibroscan for those with indeterminate FIB-4 (Step 4), and subsequent recommended management. The NCCP has face and content validity based on consensus of multiple stakeholders including VA clinicians, and high efficacy in the investigator's preliminary data. The investigators propose to adapt the multicomponent NCCP intervention for use in VA primary care and prospectively test its effectiveness for identification and severity stratification of patients with NAFLD. The investigator's approach is consistent with VA strategic priorities to implement a more "Veteran-centered" approach that improves access to care.

Innovation & Impact: This is the first study to examine the effectiveness of any NAFLD clinical care pathway in a VA primary care practice. The design is a cluster-randomized controlled trial with randomization at the level of Patient Aligned Care Teams (PACTs) in primary care, and a state-of-the-art technique to diagnose NAFLD and stage the severity of hepatic fibrosis. The investigator's formative and summative evaluation will provide key information about the feasibility, acceptability and determinants of implementation. The NCCP intervention is a paradigm shift in NAFLD care from haphazard and sporadic care into a systematic, equitable, and evidence-based approach.

Specific Aims: Aim 1. Conduct a formative evaluation to assess feasibility and acceptability of the NCCP among patients and providers; adapt the NCCP for prospective testing based on feedback. Aim 2. Examine the effectiveness of the NCCP intervention compared to usual care in improving NAFLD care processes and patient outcomes. Aim 3. Conduct a summative evaluation to identify patient and provider characteristics associated with effectiveness of NCCP and to assess future implementation. The investigator's hypothesis is that NCCP when adapted to Patient Aligned Care Teams (PACTs) in VA primary care considerably increases the identification of patients with NAFLD and those with high-risk NAFLD, and results in an increase in guideline-concordant management.

Methodology: The study will be conducted in primary care settings in a single large VA Medical Center. The investigators will conduct patient interviews and focus groups with PACTs to inform adaption of the NCCP. The investigators will then conduct a cluster-randomized trial of 16 PACTs in primary care to compare the effectiveness of NCCP to usual care in improving NAFLD care, with PACTs as unit of randomization and patients as the unit of analysis. The multicomponent intervention includes an e-trigger to identify patients eligible for NAFLD screening and calculate fibrosis scores, a structured provider education on NAFLD management and treatment recommendations, and coordination by an inter-professional team. The primary outcome will be a composite binary variable consisting of NAFLD diagnosis and risk stratification. Secondary outcomes include referral to a weight loss program, referral of patients with advanced fibrosis to hepatology specialty care, and enrollment among those referred to weight loss and hepatology specialty care. Summative evaluation will inform future implementation.

Next Steps/Implementation: The investigators study will provide information needed to support future projects to implement the NCCP in VA primary care settings. The study will also lay the foundation for a subsequent project to examine the adopted intervention's effect on weight loss and NAFLD biomarkers in patients with high-risk NAFLD.

ELIGIBILITY:
Inclusion Criteria:

Patient Aligned Care Teams (PACT) at the Michael E. DeBakey VA Medical Center

Exclusion Criteria:

* The investigators will exclude PACTs with unstable leadership (i.e., pending departure, vacancy) at time of randomization.
* PACTs participating in the focus groups in Aim 1 will be excluded in Aim 2 to avoid cross contamination.
* PACTs meeting the following criteria will be excluded from randomization in Aim 2:

  * PACTs who do not treat NAFLD,
  * PACTs not located at the main hospital,
  * PACTs with less than 100 visits within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-11-13 (Estimated)

PRIMARY OUTCOMES:
NAFLD Diagnosis and risk stratification | Baseline, 6 months
  The investigators will use chart reviews to extract unstructured data regarding the primary outcome measure: existence of EHR progress note documenting a new NAFLD diagnosis AND complete risk stratification of NAFLD (i.e., fibrosis). The investigators will use our validated process to guide uniform abstraction and classification.

SECONDARY OUTCOMES:
Fibroscan Test | Baseline, 6 & 12 months
  The investigators will extract from the EHR if a patient had a fibroscan test.
Referral to hepatology | Baseline, 6 and 12 months
  The investigators will extract from the EHR if a patient was referred to a hepatology clinic.
Hepatology Clinic Visit | Baseline, 6 and 12 months
  The investigators will extract from the EHR if a patient was seen in a hepatology clinic.
NAFLD discussion | 6 and 12 months
  The investigators will extract from the patient chart if the provider documented a discussion about NAFLD with the patient.
Referral to weight loss services | Baseline, 6 and 12 months
  The investigators will extract from the EHR if a patient was referred to weight loss services.
Enrollment in weight loss services | Baseline, 6 and 12 months
  The investigators will extract from the EHR if a patient was referred to weight loss services.

CONTACTS AND LOCATIONS:
Overall Officials: Hashem B. El-Serag, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will not share data at the individual level, only in aggregate. No data will leave the VA.

REFERENCES:
- [Derived] Godwin KM, Grigoryan L, Thrift AP, Duong H, Kanwal F, Giardina T, Kadiyala H, Zimolzak A, Patidar KR, El-Serag HB. A cluster randomized trial of a Multicomponent Clinical Care Pathway (MCCP) to improve MASLD diagnosis and management in primary care: study protocol. BMC Health Serv Res. 2025 May 6;25(1):645. doi: 10.1186/s12913-025-12737-2. PMID 40325466